CLINICAL TRIAL: NCT01756287
Title: A Randomized Controlled Trial to Alter Ocular Accommodation in Myopic Teenager With Chinese Ocular Exercise
Brief Title: Efficacy of Chinese Ocular Exercise on Visual Acuity and Ocular Accommodation in Myopic Teenager
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Shi-Ming Li, Dr., Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011CB504601
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standardized Chinese ocular exercise (Experimental): The participants are trained with standardized Chinese ocular exercise which contains accurate positions of acupuncture points and appropriate pressure on the points.
  Interventions: Other: Chinese ocular exercise
- Nonstandardized ocular exercise (Sham Comparator): The participants are trained with nonstandardized ocular exercise performed on wrong positions where no acupuncture points at all.
  Interventions: Other: Chinese ocular exercise
- Eye closure (No Intervention): The participants are told to close eyes and don't do ocular exercise at all.

INTERVENTIONS:
Other: Chinese ocular exercise — A kind of massage around the acupuncture points around the eye.
  Arms: Nonstandardized ocular exercise; Standardized Chinese ocular exercise

SUMMARY:
To assess whether Chinese ocular exercise is effective in altering distant and near visual acuity, ocular accommodation and visual symptoms in myopic teenager, and thus might have the possibility of slowing myopia progression in teenager through a weak but long-term effect.

DETAILED DESCRIPTION:
Myopia is a public health problem worldwide, especially in some Asian countries like China, Singapore, and Japan. Chinese ocular exercise, originating in 1963 with the theory of Traditional Chinese Medicine, is a kind of massage on acupuncture points around the eye to prevent myopia and alleviate visual fatigue. The exercise has been spread as a community ritual and living habit of primary and high school students for nearly half a century. However, the prevalence of myopia in Chinese children increased remarkably in recent years. Therefore, the efficacy of Chinese ocular exercise on preventing myopia or alleviating visual fatigue is widely questioned. Evidence from clinical trials of high level is needed to clarify that whether Chinese ocular exercise is effective in slowing and preventing myopia progression, or at least in part in easing the symptoms related to myopia and visual fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Visual acuity: 20/20 or better in each eye;
2. Spherical error ranging from +0.5 D to -6.0 D and astigmatism less than 1.5 D in each eye, anisometropia less than 1.0 D between the two eyes Contact lens
3. No strabismus, amblyopia and any other ocular or systematic diseases that may affect refractive development

Exclusion Criteria:

1. Currently using other interventions to control myopia progression (acupuncture, massage, drugs, ear needles and so on)
2. Unable to cooperate with the ocular examination and questionnaire survey

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Distant and near visual acuity | Before and after the intervention immediately, about 5 minutes

SECONDARY OUTCOMES:
Ocular accommodation | Before and after the intervention immediately, about 5 minutes

OTHER OUTCOMES:
Self evaluation of the improvement after the intervention | Before and after the intervention immediately, about 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ningli Wang, MD, PhD, Principal Investigator — Beijing Tongren Eye Center, Beijing Tongren Hospital, Capital Medical University, Beijing, China
Locations (1):
- Shi-Ming Li, Anyang, Henan, China

REFERENCES:
- [Derived] Li SM, Kang MT, Peng XX, Li SY, Wang Y, Li L, Yu J, Qiu LX, Sun YY, Liu LR, Li H, Sun X, Millodot M, Wang N. Efficacy of Chinese eye exercises on reducing accommodative lag in school-aged children: a randomized controlled trial. PLoS One. 2015 Mar 5;10(3):e0117552. doi: 10.1371/journal.pone.0117552. eCollection 2015. PMID 25742161